CLINICAL TRIAL: NCT03688854
Title: Effects of Short Chain Fatty Acids on Affective Processes in Humans
Brief Title: The Role of Short Chain Fatty Acids in Microbiota-gut-brain Axis
Acronym: SCFA-AP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Prof. Dr. Kristin Verbeke, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: S60501
Record Dates: First submitted 2018-09-23; First posted 2018-09-28 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Emotions; Stress; Fear

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo are capsules containing cellulose.
  Interventions: Dietary Supplement: SCFA mixture
- SCFA mixture low dose (Experimental): Encapsulated SCFA mixture in the ratio of 67:6:27 (acetate, propionate, butyrate) equivalent of 10 grams of fiber.
  Interventions: Dietary Supplement: SCFA mixture
- SCFA mixture high dose (Experimental): Encapsulated SCFA mixture in the ratio of 67:6:27 (acetate, propionate, butyrate) equivalent of 20 grams of fiber.
  Interventions: Dietary Supplement: SCFA mixture

INTERVENTIONS:
Dietary Supplement: SCFA mixture — Intracolonic administration

SUMMARY:
The role of short chain fatty acids (SCFA) in the microbiota-gut-brain axis is examined in a sample of healthy volunteers. SCFA are the major products of bacterial fermentation of dietary fiber in the colon, and are hypothesised to mediate the bidrectional communication between the gut and the residing microbiota on the one hand, and the central nervous system on the other hand. We perform a 1-week intervention with SCFA and measure their effects on a range of affective outcomes in healthy male volunteers.

DETAILED DESCRIPTION:
The study is an interventional double-blind, placebo-controlled, parallel group design with 3 arms (placebo, high-dose of SCFA, and low-dose of SCFA). The high and low doses of SCFA are equivalent to 20 and 10 grams of fiber respectively. Healthy male participants follow a low-fiber diet for the study duration (11 days). On day 4, baseline measurements are taken in the lab, including biological samples and psychophysiological measurements. Participants then consume placebo or SCFA for one week and revisit the lab on day 11 for a second measurement of the outcomes of interest. Specifically, we investigate the effect of SCFA supplementation on affective processing, including stress sensitivity, fear-related processes (e.g. extinction learning), and attentional bias to emotional stimuli. Volunteers also respond to questionnaires in relation to mood, and provide biological samples (blood and faecal samples) for analysis of circulating short chain fatty acids and microbiota composition, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Male participants
* Age range 20-40 years
* BMI range 18.5-27
* Dutch as native-language

Exclusion Criteria:

* previous or current neurological, psychiatric, gastrointestinal or endocrine disorders, or other relevant medical history
* current or recent regular medication use
* previous or current substance/alcohol dependence or abuse (> 2 units per day/14 units per week)
* one or more diagnoses based on the mini-international neuropsychiatric interview
* smoking
* night-shift work
* adherence to vegan or vegetarian diets
* use of pre- or probiotics within one month preceding the study
* use of antibiotics within 3 months preceding the study
* previous experience with one of the tasks used in the study

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Stress sensitivity | 1 year
  Induction of cognitive, physical, and social stress using Maastricht Acute Stress Test. Stress hormone cortisol is quantified.

SECONDARY OUTCOMES:
Stress sensitivity (subjective) | 1 year
  Induction of cognitive, physical, and social stress using Maastricht Acute Stress Test. Participant rate how much stress, discomfort, and pain they feel on a 10-cm visual analogue scale, with higher values indicating greater stress, discomfort, and pain. This is done prior to stress induction, in the middle, and at the end.
Cortisol awakening response | 1 year
  Measuring chronic stress by quantifying cortisol in morning samples (5 samples taken form the moment of waking every 15 minutes for 1 hour)
Fear | 1 year
  Exploring fear-related processes (conditioning, extinction, recall, and renewal) by means of a computerised task. Fear response is measured using skin conductance.
Fear (subjective) | 1 year
  Exploring fear-related processes (conditioning, extinction, recall, and renewal) by means of a computerised task. Fear response is measured subjective reports.
Attentional bias to emotional stimuli | 1 year
  Use of a dot-probe task to task attentional bias and change in attentional bias following SCFA vs. placebo supplementation. This is done via a computerised task, where reaction times are quantified.
Perceived Stress Scale (PSS) | 1 year
  The Perceived Stress Scale (PSS) was devised by Cohen et al. (1983). It is a 14-item instrument designed to measure the degree to which situations in one's life are appraised as stressful. It provides a tool for examining issues about the role of appraised stress levels in the aetiology of disease and behavioural disorders. The scale is designed such that it asks the respondent to rate the frequency of his/her feelings and thoughts related to events and situations that occurred over a selected time-frame. Notably, high PSS scores have been correlated with higher biomarkers of stress, such as cortisol.
Positive and Negative Affect Schedule (PANAS) | 1 year
  The PANAS consists of two 10-item mood scales and was developed to provide brief measures of negative affect (NA) and positive affect (PA). NA and PA reflect dispositional dimensions, with high-NA epitomized by subjective distress and unpleasurable engagement, and low-NA by the absence of these feelings. By contrast, PA represents the extent to which an individual experiences pleasurable engagement with the environment. Respondents are asked to rate the extent to which they have experienced each particular emotion within a specified time period, on a 5-point scale. The scale points are: 1 'very slightly or not at all', 2 'a little', 3 'moderately', 4 'quite a bit', and 5 'very much'.
Depression, Anxiety, and Stress Scale (DASS-21) | 1 year
  The DASS is a set of three self-report scales designed to measure the negative emotional states of depression, anxiety and stress. Each of the three DASS scales contains 14 items, divided into subscales of 2-5 items with similar content. The Depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest/involvement, anhedonia, and inertia. The Anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The Stress scale is sensitive to levels of chronic non-specific arousal. Subjects are asked to use 4-point severity/frequency scales to rate the extent to which they have experienced each state over the past week. Scores for Depression, Anxiety and Stress are calculated by summing the scores for the relevant items. DASS21 will be used in the present study.
Gastointestinal symptom rating scale (GSRS) | 1 year
  The GSRS (Svellund et al., 1988) is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms. The reliability and validity of the GSRS are well-documented, and norm values for a general population are available.
Microbiota composition | 1 year
  Analysis of microbiota composition at baseline and after SCFA mixture administration in faecal samples
Circulating SCFA | 1 year
  Measurement of SCFA concentration in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Verbeke, Prof, Principal Investigator — KU Leuven
Locations (1):
- UZ Leuven/Stresslab, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided